CLINICAL TRIAL: NCT06596018
Title: Efficacy and Safety Evaluation of Combined Preoperative Radiotherapy in Breast Cancer Patients With No Response to Initial Neoadjuvant Chemotherapy
Brief Title: Assessing Combined SBRT in Breast Cancer Non-Responders to Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y2024-0756
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-09

CONDITIONS: Breast Adenocarcinoma
Keywords: breast cancer; chemo-resistance; neoadjuvant radiation; pCR rate
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Active Comparator): Patients in this group will continue to follow the original chemotherapy using anthracycline and/or taxane based regimens, according to their physician's preference and center policy
  Interventions: Drug: Chemotherapy
- The SBRT-combined group (Experimental): The intervention group will receive SBRT treatment. The specific plan for SBRT is to target the primary tumor region with 24Gy/3. After the completion of SBRT, patients will continue the remaining courses of neoadjuvant chemotherapy.
  Interventions: Radiation: SBRT; Drug: Chemotherapy

INTERVENTIONS:
Radiation: SBRT — Target the primary tumor region with a single dose of 8Gy using 6MV-X rays, administered once a day for three consecutive days.
  Arms: The SBRT-combined group
Drug: Chemotherapy — Continue to follow the original chemotherapy regimen（anthracycline and/or taxane based regimens）

SUMMARY:
The goal of this clinical trial is to assess whether the addition of preoperative stereotactic body radiation therapy (SBRT) can improve pathological complete response (pCR) rates and safety in breast cancer patients who do not respond to initial neoadjuvant chemotherapy. The main questions it aims to answer are:

* Can the combination of SBRT with chemotherapy increase pCR rates in non-responders to initial neoadjuvant chemotherapy?
* Does the addition of SBRT to chemotherapy have acceptable safety and tolerability profiles?

Participants in this trial will be early or locally advanced breast cancer patients who have shown no response to two cycles of standard neoadjuvant chemotherapy. They will be randomly assigned to either continue with the standard chemotherapy (control group) or receive SBRT in addition to continuing the standard chemotherapy (intervention group). The primary outcome measures will be pCR rate and breast conservation rate. Secondary outcomes will include 3-year local progression-free survival, overall survival, surgical complications, and treatment toxicities.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy is a crucial component in the comprehensive treatment of breast cancer patients, particularly for those with large initial tumors, axillary lymph node metastasis, HER-2 positive, or triple-negative disease. However, some patients do not achieve the desired pathological complete response (pCR) after neoadjuvant chemotherapy. The CTNeoBC meta-analysis has shown that breast cancer patients who achieve pCR after neoadjuvant therapy have a better prognosis compared to those who do not. Specifically, patients who reach pCR exhibit a recurrence rate of less than 10%, whereas those who fail to achieve pCR may have a recurrence rate as high as 50%. On the other hand, in breast-conserving therapy, patients typically undergo boost radiotherapy targeted at the tumor bed, which is administered after the completion of whole-breast radiotherapy. Existing evidence suggests that advancing the radiotherapy boost to the preoperative period is equally effective and safe. To enhance the treatment outcomes for patients who do not respond to initial standard chemotherapy, the investigators have designed this prospective preliminary study to assess the efficacy and safety of stereotactic body radiation therapy (SBRT) when added to neoadjuvant therapy in this population of chemotherapy non-responders.

This study is a prospective, randomized controlled trial. Patients first undergo standard neoadjuvant chemotherapy, with tumor size evaluated through physical examination or ultrasound after each cycle, and breast MRI for tumor assessment after two cycles. Patients who are assessed as having stable disease (SD) or progressive disease (PD) according to RECIST criteria are considered non-responders to initial neoadjuvant chemotherapy. Participants will be randomly allocated in a 1:1 ratio to either the control group or the intervention group. The control group will continue to follow the original chemotherapy regimen, while the intervention group will receive SBRT treatment. The specific plan for SBRT is to target the primary tumor region with a single dose of 8Gy using 6MV-X rays, administered once a day for three consecutive days. After the completion of SBRT, patients will continue the remaining courses of neoadjuvant chemotherapy. Both groups of patients will subsequently undergo standard surgery based on efficacy assessment, followed by whole-breast hypofractionated radiotherapy 4-6 weeks postoperatively, with a plan of 40-42.5Gy/15-16 fractions, without a boost to the original tumor area.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histologic diagnosis of invasive adenocarcinoma of the breast;
* Stage T1-4N+M0 breast cancer (i.e., stages II and III);
* Breast MRI showing no extracapsular extension of lymph node involvement;
* The standard neoadjuvant chemotherapy regimen has been deemed ineffective after two cycles, with disease assessed as stable (SD) or progressive (PD) according to RECIST 1.1 criteria;
* ECOG performance status score of 0-2;
* Screening laboratory values must meet the following criteria:

  i. White blood cells (WBCs) ≥ 2000/μL ii. Absolute neutrophil count (ANC) ≥ 1500/μL iii. Platelets ≥ 100 x 103/μL iv. Hemoglobin ≥ 11.0 g/dL v. Serum creatinine ≤ 2 mg/dL (or glomerular filtration rate ≥ 40 ml/min) vi. AST ≤ 2.5 x upper limit of normal (ULN) vii. ALT ≤ 2.5 x ULN viii. Total bilirubin within normal limits (except subjects with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL) ix. INR ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulant(s) x. Negative HIV screening test xi. Negative screening tests for Hepatitis B and Hepatitis C. Patients with positive results that do not indicate true active or chronic infection may enroll after discussion and consensus agreement by the treating physician and principal investigator.

Exclusion Criteria:

* Evidence of metastatic disease;
* Known additional malignancy that is progressing or has required active treatment within the past 3 years；
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug；
* Patients with other concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study；
* Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Breast conservation rate | Intraoperative
  Breast conservation rate
pCR rate | At the end of chemotherapy up to 21 weeks
  Pathological complete response (pCR), defined by the absence of invasive residual primary tumor in the breast and lymph node.The primary objective of this study is to compare pCR rates after continuing chemotherapy plus SBRT versus continuing chemotherapy alone in patients with non-response to initial 2 cycles of neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
3-year PFS | 3 years after completion of treatment
  PFS is a measure of the time from the start of treatment until the disease progresses or a recurrence is observed, or until death occurs from any cause.
Acute and late toxicities | At the end of chemotherapy and after surgery and after radiotherapy At the end of chemotherapy and after surgery and after radiotherapy: up to 30 weeks
  Acute and late toxicities (CTCAE v 4.0)

CONTACTS AND LOCATIONS:
Locations (1):
- The Department of Radiation Oncology，the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided